CLINICAL TRIAL: NCT05782764
Title: A Single-arm, Exploratory Clinical Study of 3-day Continuous Intravenous Pump of Endostatin (Endostar) Combined With Chemotherapy and Immune Checkpoint Inhibitor in the Treatment of Advanced Lung Squamous Cell Carcinom
Brief Title: A Study of Endostar Combined With Chemotherapy and Immunotherapy in Lung Squamous Cell Carcinom
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Xichao Dai, Yancheng Clinical College, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-003
Record Dates: First submitted 2023-03-04; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Lung Squamous Cell Carcinoma
MeSH Terms: interventions — endostar protein; Drug Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Recombinant human endostatin (CIV72h, D1-D3, 14 tubes) was administered by continuous intravenous infusion every 3 weeks. The drug was discontinued until disease progression or intolerable side effects.
  Interventions: Drug: To explore the efficacy and safety of immune checkpoint inhibitor combined with endostar and chemotherapy in the treatment of advanced lung squamous cell carcinoma (stage IIIB-IV).

INTERVENTIONS:
Drug: To explore the efficacy and safety of immune checkpoint inhibitor combined with endostar and chemotherapy in the treatment of advanced lung squamous cell carcinoma (stage IIIB-IV). — immune checkpoint inhibitor combined with endostar and chemotherapy in the treatment of advanced lung squamous cell carcinoma (stage IIIB-IV).
  Other Names: Endostar combined with immune checkpoint inhibitor and chemotherapy in the treatment of advanced lung squamous cell carcinoma (stage IIIB-IV)

SUMMARY:
To explore the efficacy and safety of immune checkpoint inhibitor combined with endostar and chemotherapy in the treatment of advanced lung squamous cell carcinoma (stage IIIB-IV).

DETAILED DESCRIPTION:
This study is a prospective, single-arm, single-center phase II study to evaluate the efficacy and safety of immune checkpoint inhibitors in combination with chemotherapy and recombinant human endostatin in patients with advanced (stage IIIB-IV) squamous non-small cell lung cancer. Patients with locally advanced stage ⅢB/ⅢC, metastatic or recurrent stage IV squamous NSCLC who were not operable and could not receive radical concurrent chemoradiotherapy were selected after signing informed consent. Eligible subjects who met the inclusion criteria were screened for immune checkpoint inhibitor combined with chemotherapy and recombinant human endostatin. After cycles 4 to 6, maintenance therapy with an immune checkpoint inhibitor and endostatin was administered until disease progression, unacceptable toxicity, withdrawal of consent, initiation of additional antineoplastic therapy, death, or other protocol-specified discontinuation of treatment, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provided written informed consent before performing any trial-related procedures;

  2. Aged from 18 to 75 years old (including 75 years old);

  3. Patients with histologically or cytologically confirmed, locally advanced (stage IIIB/IIIC), metastatic, or recurrent (stage IV) squamous NSCLC according to the International Association for the Study of Lung Cancer and American Joint Committee on Classification of Cancer 8th Edition TNM classification of Lung cancer, who are inoperable and not amenable to definitive concurrent chemoradiotherapy;

  4. At least one radiographic measurable lesion according to response evaluation Criteria in Solid Tumors (RECIST, version 1.1);

Exclusion Criteria:

1. If the tumor had invaded large blood vessels on imaging (CT or MRI), or it was judged that the tumor was likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study;
2. Currently participating in an interventional clinical study treatment or receiving another study drug or study device within 4 weeks before the first dose;
3. Presence of active hemoptysis, active diverticulitis, abdominal abscess, gastrointestinal obstruction, and peritoneal metastasis requiring clinical intervention;
4. Grade III-IV congestive heart failure (New York Heart Association class) with poorly controlled clinically significant arrhythmias;
5. Any arterial thrombosis, embolism, or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, occurred within 6 months before enrollment;
6. Known allergic reactions to the study drugs;
7. Patients requiring long-term systemic corticosteroids. Patients who required intermittent use of bronchodilators, inhaled corticosteroids, or topical corticosteroid injections due to COPD or asthma were eligible.
8. Symptomatic central nervous system metastases Patients with asymptomatic brain metastases or symptomatic stabilization of treated brain metastases were eligible to participate in the study if they met all the following criteria: measurable disease outside the central nervous system; No metastasis was found in midbrain, pons, cerebellum, meninges, medulla oblongata or spinal cord. Maintain a clinically stable state for at least 2 weeks; Hormone therapy was stopped 3 days before the first dose of study drug;
9. Active infection requiring treatment or use of systemic anti-infective agents within 1 week before the first dose;
10. Has not fully recovered from any intervention-related toxicity and/or complications before starting treatment (i.e., grade ≤1 or baseline, excluding fatigue or alopecia);
11. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive);
12. Untreated active hepatitis B (defined as both HBsAg positivity and HBV-DNA copies greater than the upper limit of normal in the laboratory of the participating center);

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2months ~ 10 months
  Progression-free survival time
ORR | about 10months
  objective response rate
AE | about 10months
  adverse reactions

SECONDARY OUTCOMES:
OS | about 30 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xichao Dai, Principal Investigator — Yancheng Clinical College of Xuzhou Medical University
Locations (1):
- Yancheng Clinical College of Xuzhou Medical University, Yancheng, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No